CLINICAL TRIAL: NCT01449305
Title: Research on Effectiveness of Nanoone Woman Underwear Using in the Management of Dysmenorrhea
Brief Title: Effectiveness of Nanoone Woman Underwear Using in the Management of Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Yi Enterprise, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Nanoone
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2011-08

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

ARMS (1):
- Nanoone Woman Underwear (Experimental): "Nanoone" negative ion of textiles, which is health material specifically designed for human body, in short distance and long time to produce negative ion, the human body really needed, it can neutralize free radical in the human body.
  Interventions: Device: Nanoone Woman Underwear

INTERVENTIONS:
Device: Nanoone Woman Underwear — Chen Yi Enterprise, Co., Ltd. design a kind of negative ion materials can supply delocalized electron, and add fiber inside, make clothes to wear in the body, no external power or battery, only depend on infrared body photon hit of thermoelectric effect or heart compression pulse, blood flow of piezoelectric, therefore can sustained sufficient amount of effective negative ion, to eliminate positive ions in vivo, or make oxygen free radical to obtain the lack electrons. Decrease active free radical and get non toxic effect in short time.

SUMMARY:
To evaluate the mean change in menstrual pain intensity during menstrual cycles from baseline after wearing Nanoone Woman Underwear in women with primary dysmenorrhea

DETAILED DESCRIPTION:
The severity of dysmenorrhea pain experienced by subjects will be evaluated on a VAS, ranging from zero (no pain) to ten (very severe pain). Subjects will be asked to use the VAS scoring system to record, on a provided sheet, their experienced menstrual pain level daily during menstrual bleeding for a total of three consecutive menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged below 40 years old.
2. Screened by inquiry and diagnosed as primary dysmenorrhea by gynaecologist with pelvic ultrasonography.
3. Female subject who is:

   * using adequate contraception since last menstruation and no plan for conception during the study.
   * non-lactating.
   * has negative pregnancy test (urine) within 14 days prior to the study.
4. Informed consent form signed.

Exclusion Criteria:

1. Sensitivity to study product.
2. Patient has been diagnosed with secondary dysmenorrhea (defined as identifiable pelvic pathology).
3. Patient has clinically significant physical disability or abnormal findings on physical examination or laboratory testing judged by the investigator or co-investigator.
4. Participation of any clinical investigation during the last 30 days.

Ages: 13 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PingTung Christian Hospital, Pingtung City, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-four (44) subjects enrolled into the study. Forty-two (42) subjects completed the study from 2011-10-11 to 2012-06-23 at the PingTung Christian Hospital (60, Dallan Road, Pingtung, Taiwan).
Pre-assignment Details: This is an Open-label study design. The subject must be qualified for the study by fulfilling all of the inclusion and none of the exclusion criteria. Laboratory values which are out of reference range will not qualify unless the physician deems the deviation not clinically significant (NCS).
Groups:
- Nanoone Woman Underwear: "Nanoone" negative ion of textiles, which is health material specifically designed for human body, in short distance and long time to produce negative ion, the human body really needed, it can neutralize free radical in the human body. The subjects were required to wear the Nanoone Woman Underwear during each menstrual cycle for a total of three consecutive menstrual cycles.
Period: Overall Study
Arm/Group | Nanoone Woman Underwear
Started | 44
Completed | 42
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nanoone Woman Underwear
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 41
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 44

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change in Maximum Pain Level at Each Menstrual Cycle From Baseline
Description: The severity of dysmenorrhea pain experienced by subjects will be evaluated on a VAS, ranging from zero (no pain) to ten (very severe pain).
Time Frame: baseline, first menstrual cycle, second menstrual cycle and third menstrual cycle
Population: Subjects were asked to use the VAS scoring system to record, on a provided sheet, their experienced menstrual pain level daily during menstrual bleeding for a total of three consecutive menstrual cycles in house. Primary objective was analyzed based on the Per-protocol (PP) population.
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Nanoone Woman Underwear
Number analyzed (Participants) | 42
scores
  First menstrual cycle | -0.810 (2.04)
  Second menstrual cycle | -1.29 (1.81)
  Third menstrual cycle | -1.74 (2.24)

2. Other Pre Specified Outcome: Medicine Administration for Pain Relief During Study Period
Description: Continue taking pharmacological pain relief if required for subjects was allowed during study period, and it had been recorded.
Time Frame: first menstrual cycle, second menstrual cycle and third menstrual cycle
Population: It was analyzed based on the PP population.
Measure: Number; unit: percentage of participants
Arm/Group | Nanoone Woman Underwear
Number analyzed (Participants) | 42
percentage of participants
  First menstrual cycle | 21.4
  Second menstrual cycle | 9.52
  Third menstrual cycle | 7.14

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Nanoone Woman Underwear
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No